CLINICAL TRIAL: NCT00637338
Title: A Phase 1, Randomized, Placebo-Controlled, Sequential Parallel Group, Multiple Dose Escalation Trial To Evaluate The Safety, Tolerability, Pharmacokinetics, And Pharmacodynamics Of 4, Once-Weekly Subcutaneous Doses Of PF-04603629 To Subjects With Type 2 Diabetes Mellitus
Brief Title: Multiple Dose Escalation Trial Of PF-04603629 Given To Subjects With Type 2 Diabetes Mellitus
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: B0571002
Record Dates: First submitted 2008-03-10; First posted 2008-03-17 (Estimated); Last update posted 2009-07-31 (Estimated); Status verified 2008-11

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Long-acting GLP-1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — PF 04603629

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- PF-04603629 (Experimental): The dose range initially planned is 3 mg up to 70 mg, although the specific doses administered may be modified based on emerging study data.
  Interventions: Biological: PF-04603629
- Placebo (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: PF-04603629 — Subjects will be given either PF-04603629 or Placebo in a blinded fashion. Subjects will receive 4 weekly injections of PF-04603629 or Placebo.
  Arms: PF-04603629
Biological: Placebo — Subjects will be given either PF-04603629 or Placebo in a blinded fashion during the study. Subjects will receive 4 weekly injections of PF-04603629 or Placebo.
  Arms: Placebo

SUMMARY:
PF-04603629 is being investigated for the treatment of Type 2 diabetes mellitus (T2DM). Specifically, PF-04603629 is a protein that is a combination of exendin-4 (a glucagon-like peptide-1 (GLP-1) mimetic currently marketed as Byetta®) fused to human transferrin (a naturally occuring protein) in order to increase the concentration of exendin-4 in the blood. The purpose of this study is to characterize the safety, tolerability, pharmacokinetics, and pharmacodynamics of PF-04603629 following multiple escalating subcutaneous doses in adult subjects with T2DM.

DETAILED DESCRIPTION:
B0571002 was terminated August 19 2008 due to the decision to discontinue development of PF-04603629 after observing (in both B0571001 and B0571002) a trend for a reversible increase in heart rate within the normal range, which occurred at efficacious doses. Thus, the compound was primarily terminated due to safety concerns, although there was no immediate safety risk to any subject in the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 2 diabetes mellitus who are not taking any treatment or are taking metformin (with no change in the treatment, including dose, over the past 2 months). Subjects previously treated with a sulfonylurea in combination with metformin may be eligible if switched over to metformin only for a minimum of 4 weeks before dosing.
* Male and/or female subjects (females will be women of non-childbearing potential) between the ages of 18 and 70 years, inclusive.
* Body Mass Index (BMI) of approximately 22 to 40 kg/m2
* Fasting C-peptide test result must be >0.4 nmol/L.
* HbA1c ≥7% and ≤11%. If the subject requires to be washed off a sulfonylurea, the HbA1c limits will be ≥7% and ≤9.5%.

Exclusion Criteria:

* Screening fasting blood glucose, ≤60 or ≥270 mg/dL. One repeat screening fasting blood glucose will be allowed.
* Previous treatment with an approved or investigational GLP-1 mimetic.
* Have a known allergy to yeast, yeast-derived or yeast containing products.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2008-04; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
To characterize the pharmacokinetics of PF-04603629 in serum after administration of escalating, multiple, subcutaneously injected doses of PF-04603629 to subjects with T2DM. | 4 weeks per dose group
To evaluate the effects of multiple, escalating, subcutaneously injected doses of PF-04603629, on the pharmacodynamic responses of glucose, insulin, C-peptide and glucagon during a mixed meal tolerance test (MMTT). | 4 weeks per dose group
To describe the safety and tolerability of escalating, multiple, subcutaneously injected doses of PF-04603629 administered to subjects with T2DM. | 4 weeks per dose group

SECONDARY OUTCOMES:
To evaluate the effect of multiple, escalating, subcutaneously injected doses of PF-04603926 on additional exploratory efficacy biomarkers related to this drug's target in subjects with T2DM. | 4 weeks per dose group

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (4):
- United States (4):
  - Pfizer Investigational Site, Phoenix, Arizona
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, Wichita, Kansas
  - Pfizer Investigational Site, Portland, Oregon

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B0571002&StudyName=Multiple%20Dose%20Escalation%20Trial%20Of%20PF-04603629%20Given%20To%20Subjects%20With%20Type%202%20Diabetes%20Mellitus